CLINICAL TRIAL: NCT05159687
Title: A Randomized, Prospective, Placebo-Controlled, Crossover Study of Atomoxetine in the Prevention of Vasovagal Syncope (POST7)
Brief Title: Study of Atomoxetine in the Prevention of Vasovagal Syncope
Acronym: POST7
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POST 7
Record Dates: First submitted 2021-11-02; First posted 2021-12-16 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Vasovagal Syncope
Keywords: reflex fainting; vasovagal syncope; randomized clinical trial; quality of life; Atomoxetine
MeSH Terms: conditions — Syncope, Vasovagal | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atomoxetine (Active Comparator): Atomoxetine 40 mg PO BID (morning and late afternoon) Dosing will start at 40 mg daily for 3 days1 week, followed by a forced titration to 40 mg BID, as per the FDA label for atomoxetine.
  Interventions: Drug: Atomoxetine Hydrochloride
- Placebo (Placebo Comparator): Matching placebo will be identical in appearance to the active treatment pill. BID (morning and late afternoon)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride — Atomoxetine 40 mg PO BID (morning and late afternoon) Dosing will start at 40 mg daily for 3 days1 week, followed by a forced titration to 40 mg BID, as per the FDA label for atomoxetine
  Arms: Atomoxetine
Drug: Placebo — Placebo Comparator: Placebo Matching placebo will be identical in appearance to the active treatment pill. BID (morning and late afternoon)
  Arms: Placebo

SUMMARY:
Project rationale: Vasovagal syncope (VVS) affects up to 50% of people, and recurrent syncope markedly reduces quality of life. We recently reported that it is frequently associated with injury and not surprisingly with clinical anxiety. Although conservative measures help many patients there remain many who require more care. CIHR-funded studies have shown that fludrocortisone and midodrine are effective but cannot be used in patients with contraindications such as hypertension and heart failure. Pacemakers are partially effective in older patients, but this is established only in the small minority with proven asystole. There remains a need for a simple, once-daily medication with few contraindications that can be used as first-line therapy for most patients with recurrent vasovagal syncope.

Preliminary Studies: Norepinephrine transport (NET) inhibitors show promise as a novel treatment. Three (reboxetine, sibutramine, and atomoxetine) all prevent vasovagal syncope in healthy subjects and vasovagal syncope patients on tilt tests. Atomoxetine, approved to treat attention deficit disorder, is a highly selective NET inhibitor. We reported a proof-of-principle, randomized, placebo-controlled trial of the efficacy of atomoxetine to prevent vasovagal syncope on tilt table tests. Patients underwent tilt testing after receiving either atomoxetine 40 mg or placebo. Fewer VVS patients fainted with atomoxetine than placebo (10/29 vs. 19/27; odds ratio 0.22, p < 0.01). Our meta-analysis of the effects of NET inhibition on the vasovagal reflex induced by tilt tests was highly positive. A pre-post study showed that sibutramine reduced syncope frequency in highly symptomatic and drug-refractory patients. A similar pre-post study showed that atomoxetine also reduces syncope frequency about 85% in patients with frequent and drug-intolerant or drug-resistant vasovagal syncope. Therefore,NET inhibition by atomoxetine merits assessment based on positive proof-of-principle studies, an apparent class effect, and two open-label pre-post studies. These results provide the rationale for a formal randomized, placebo-controlled, crossover trial of atomoxetine in moderate-to-high risk patients with VVS.

Hypothesis: We will test the hypothesis that oral atomoxetine prevents syncope in patients with recurrent VVS.

The Study: Patients will be included based on a positive Calgary Syncope Symptom Score and a history of at least 2 faints in the previous year. Eligible patients will be randomized to atomoxetine 40 mg po twice daily or matching placebo in a randomized, placebo-controlled, parallel design, double-blind, crossover trial. Each arm will last 6 months with a 1-week washout period. The primary outcome measure will be the proportion of patients with at least 1 syncope recurrence. The study will be powered to detect a beneficial odds ratio of 0.5, selected on the basis of the control outcome rates in 2 similarly designed, previous studies and international expert requirements for effect size. A sample size of 180 subjects will provide 85% power of detecting a difference between the arms at p<0.05. We will assess the effects of atomoxetine on quality of life, anxiety, injury, and the cost-effectiveness of atomoxetine treatment, and the effects of genetic factors on outcomes.

Substudies : The quality of life scales will be the SF-36 and the Euroqol EQ5D, which will also be used as the health utility index for the economic studies. The depression and anxiety scales will be the Hospital and Anxiety Depression Score (HADS) and the General Anxiety Disorder - 7 Score (GAD-7). Clinical anxiety is highly prevalent in patients with recurrent syncope. Injury will be self-reported using our published definitions. The health economic substudy will be from the health system perspective and will use Alberta administrative data. DNA will be collected from spit acquired in the Oragene saliva self-collection kits, and an initial candidate gene study might include alleles of CYP2D6, COMT, the serotonin (SLC6A4) and norepinephrine (SLC6A2) reuptake transporters, and the 5HT1A and 5HT3 receptors.

Summary: Adults who faint recurrently are highly symptomatic. There are no therapies suitable for most patients have withstood the test of randomized clinical trials. If successful, atomoxetine will reduce syncope and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Syncope according to the American College of Cardiology Guidelines 2017
2. At least 2 vasovagal syncope spells in the preceding 12 months
3. At least -2 on the Syncope Symptom Score for Structurally Normal Hearts
4. At least 18 years old with informed consent

Exclusion Criteria:

1. Other cause of syncope
2. A 5-minute stand test resulting in the diagnosis Orthostatic Hypotension or Postural Orthostatic Tachycardia Syndrome
3. An inability to give informed consent
4. Pregnant
5. Unwilling or unable to use adequate birth control while on study drug.
6. An important valvular, coronary, myocardial, or conduction abnormality, or significant arrhythmia
7. Uncontrolled hypertension
8. Uncontrolled hyperthyroidism
9. A permanent pacemaker
10. Taking or has recently taken a monoamine oxidase inhibitor
11. Pheochromocytoma
12. Glaucoma
13. Prior use of atomoxetine for syncope
14. Clinical need for atomoxetine or another potent norepinephrine transporter inhibitors (Ki NET < Ki SERT, Ki NET > 10 Ki atomoxetine),
15. Current use of β-blocker, bupropion, α1-adrenergic agonists or antagonists, tricyclic antidepressants, serotonin reuptake inhibitors, scopolamine, theophylline, or fludrocortisone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the proportion of patients having at least one syncope recurrence. | Within 12 months period of the study
  one syncope recurrence

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | every 6 months of the study up to 12 months
  The total score is out of 42, (21 per subscale). Scores are derived by summing responses for each of the two subscales or for the scale as a whole Higher scores indicate greater levels of anxiety or depression. The total HADS score may be regarded as a global measure of psychological distress
Generalized Anxiety Disorder score | every 6 months of the study up to 12 months
  The GAD-7 is useful in primary care and mental health settings as a screening tool and symptom severity measure for the four most common anxiety disorders (Generalized Anxiety Disorder, Panic Disorder, Social Phobia and PostTraumatic Stress Disorder).
  It is 70-90% sensitive and 80-90% specific across disorders / cutoffs (see Evidence section for more).
  Higher GAD-7 scores correlate with disability and functional impairment (in measures such as work productivity and health care utilization)
EQ-5D-3L | every 6 months of the study up to 12 months
  The EQ-5D-3L classification system consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each with three levels: no problems "1", moderate problems "2", and severe problems "3". Each health state is described as a vector of these five dimensions. With 3 levels for each dimension, the EQ-5D-3L describes 243 distinct health states, with 11111 being the best health state (full health), and 33333 the worst health state.
  In addition to the classification system, each of the instruments also includes a visual analogue scale (EQ VAS). The EQ VAS records the respondent's self-rated health on a visual analogue scale from 0 to 100, whereby 0 indicates 'the worst health you can imagine', and 100 'the best health you can imagine'. This information can be used as a quantitative measure of health as judged by the individual respondents.
Rand 36 Scale | every 6 months of the study up to 12 months
  The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. Aggregate scores are compiled as a percentage of the total points possible, using the RAND scoring table
ISQL form | every 6 months of the study up to 12 months
  The ISQL is a brief valid measure of the impact of syncope on quality of life. It measures impairment, fear, depression, and physical limitations, and correlates with recent syncope frequency.
Medical Utilization form | every 3 months of the study up to 12 months
  Cost, and cost-effectiveness

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandhu RK, Raj SR, Hamzeh R, Sheldon RS; POST 7 Investigators. The Seventh Prevention of Syncope Trial (POST VII)-A randomized clinical trial of atomoxetine for the prevention of vasovagal syncope: Rationale and study design. Am Heart J. 2023 Aug;262:49-54. doi: 10.1016/j.ahj.2023.04.012. Epub 2023 Apr 24. PMID 37100187